CLINICAL TRIAL: NCT01061385
Title: IDE G090121 A Prospective, Randomized Multicenter Study to Evaluate the Safety and Efficacy of the ReShape Intragastric Balloon (RIBTM) in Obese Subjects
Brief Title: The Safety and Efficacy of the ReShape Intragastric Balloon in Obese Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ReShape Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REDUCE-IDE
Record Dates: First submitted 2010-02-01; First posted 2010-02-03 (Estimated); Results first posted 2015-12-07 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ReShape Intragastric Balloon (Experimental): Patients receiving the ReShape Intragastric Balloon
  Interventions: Device: ReShape Intragastric Balloon
- Control Arm (Other): Weight loss using behavior modification (diet and exercise counseling) alone
  Interventions: Other: Control Arm

INTERVENTIONS:
Device: ReShape Intragastric Balloon — Placement of ReShape Medical Intragastric Balloon for twenty four weeks
  Arms: ReShape Intragastric Balloon
Other: Control Arm — Behavioral Modification (Diet and exercise counseling) alone
  Arms: Control Arm

SUMMARY:
The study evaluated the safety and efficacy of the ReShape Intragastric Balloon as an adjunct to diet and exercise in obese patients compared with diet and exercise alone. The study device is designed to occupy space within the stomach and induce satiety. After approval from the institutional review board, patients provided written consent and were randomized to the treatment group (with endoscopic placement of study device) or the control group (no placement of study device) on an unblinded basis. Both groups received similar diet and exercise counseling. After 24 weeks, the device was removed. Patient weight, adverse events, and quality of life data were evaluated throughout the 48 week study duration.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged ≥ 20 years and ≤ 60 years;
2. At screening, body mass index (BMI) ≥ 30 Kg/m^2 and ≤ 40 Kg/m^2;
3. Have a history of obesity (BMI ≥ 30 kg/m^2) for at least 6 months and have failed other weight-reduction alternatives, such as supervised diet, exercise and behavioral modification programs;
4. Subject is willing to commit to a long-term low calorie (1000-1500 calories/day) supervised diet;
5. Subject has reasonable weight loss expectations (accept a goal of losing up to 15% of body weight after 24 weeks);
6. At screening, total Beck Depression Inventory (BDI) score < 12 points, and BDI affective subscale score < 7 points.
7. Subject is able to follow requirements outlined in the protocol, including complying with the visit schedule, and willing to undergo protocol-specific procedures, e.g., endoscopy, local sedation, general anesthesia, electrocardiography (ECG), and/or clinical laboratory testing;
8. Subject is willing to take prescribed proton pump inhibitors (PPIs);
9. Subject is able to provide written informed consent;
10. If female of child-bearing potential, the subject is willing to use contraception (e.g., birth control pills, condoms, abstinence) and avoid pregnancy during the study.

Exclusion Criteria:

1. Participating in an organized weight loss program (e.g., Weight Watchers);
2. Parkinson's disease;
3. Chronic narcotic use;
4. Clinically relevant abdominal adhesions (e.g., history of bowel obstruction);
5. History or symptoms of gastrointestinal (GI) surgery (excluding uncomplicated appendectomy and cholecystectomy), obstruction, and/or adhesive peritonitis;
6. History or symptoms of clinically significant esophageal or GI motility disorders;
7. A hormonal or genetic cause for subject's obesity;
8. A history of myocardial infarction in the previous 6 months, current New York Heart Association (NYHA) Functional Class III or IV (heart failure) or cardiac arrhythmia (e.g., atrial fibrillation);
9. History or symptoms of varices, bowel obstruction, congenital or acquired GI anomalies (e.g., atresias, stenosis, stricture, and/or diverticula), severe renal, hepatic, and/or pulmonary disease;
10. History or symptoms of inflammatory bowel disease, such as Crohn's disease;
11. History or symptoms of uncontrolled or unstable thyroid disease;
12. Subjects with a positive breath test for Helicobacter pylori at screening;
13. History or symptoms in the past 12 months of significant irritable bowel disease, peritonitis, active esophagitis, gastric or duodenal ulceration, or GI bleeding;
14. History of esophageal and/or stomach cancer.
15. Type I diabetes;
16. Placement of previous intragastric balloon or similar device with associated adverse; or any endogastric procedure within the last 6 months;
17. Ongoing treatment with anticoagulants, steroids, aspirin (> 81 mg/day), non-steroidal anti-inflammatory drugs (NSAIDS), or other medications known to be gastric irritants or to reduce GI motility, and unwillingness to discontinue the use of these concomitant medications;
18. Concomitant use of prescription, non-prescription, or over-the-counter weight loss medications or supplements at any time during the study;
19. Evidence of untreated psychiatric or eating disorders, such as major depression, schizophrenia, substance abuse, binge eating disorder, or bulimia;
20. Pregnancy, breast feeding, or intention of becoming pregnant during the study (if female of childbearing potential);
21. Known allergy to silicone;
22. A history of anemia
23. Participation in another investigational trial within 1 month of screening or planned enrollment during the study period.
24. Presence of peptic ulcerations, hiatal hernia (> 2 cm), patulous pyloric channel, erosive esophagitis, varices, angiectasia, Barrett's esophagus or other findings deemed exclusionary in the opinion of the investigator.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-02; Primary Completion 2011-03 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Lou Mooney, Study Director — ReShape Medical

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Arm: Patients presenting for weight loss using behaviour modification (diet and exercise) alone.
  Behavioral modification: Diet and exercise
Period: Overall Study
Arm/Group | ReShape Intragastric Balloon | Control Arm
Started | 21 | 9
Completed | 20 | 8
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — subject decision not related to AE | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants meeting study inclusion/exclusion criteria
Groups:
- Total: Total of all reporting groups
Arm/Group | ReShape Intragastric Balloon | Control Arm | Total
Number analyzed (Participants) | 21 | 9 | 30
Age, Continuous [Mean (Full Range); unit: years] | 38.9 [26 to 59] | 45.3 [37 to 55] | 40.8 [26 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 9 | 26
  Male | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: %Excess Weight Loss
Description: the difference between the %EWL between treatment and control groups must be clinically significant
Time Frame: 36 Weeks
Measure: Mean (Standard Deviation); unit: percent excess weight loss
Groups:
- Control: Control subjects receiving diet and exercise counseling only
Arm/Group | ReShape Intragastric Balloon | Control
Number analyzed (Participants) | 21 | 9
percent excess weight loss | 20.2 (16.7) | 12.7 (19.3)
Statistical Analysis 1: Comparison: ReShape Intragastric Balloon vs Control; Test type: Superiority or Other; p = 0.2922, t-test, 1 sided; Mean Difference (Net) = 7.5, 95% CI 2-sided [-6.8 to 21.7]

2. Secondary Outcome: Percentage of Subjects With >=25% Excess Weight Loss (EWL)
Description: a between-group comparison of percentage of treatment subjects achieving >=25% EWL (using the Metropolitan Life Tables (ML) method) compared to the percentage of control group subjects achieving >= 25%EWL at 12 months
Time Frame: 12 months
Measure: Number; unit: percentage of subjects
Arm/Group | ReShape Intragastric Balloon | Control Arm
Number analyzed (Participants) | 20 | 8
percentage of subjects | 30 | 25
Statistical Analysis 1: Comparison: ReShape Intragastric Balloon vs Control Arm; Test type: Superiority or Other; Mean Difference (Net) = 5, 95% CI 2-sided [-37.7 to 38.0] — The 95% CI range above is calculated for the current estimated value

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | ReShape Intragastric Balloon | Control Arm
Serious Adverse Events (participants affected / at risk) | 3/21 | 0/9
Other Adverse Events (participants affected / at risk) | 21/21 | 6/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ReShape Intragastric Balloon (N=21) | Control Arm (N=9)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
periorbital edema (Eye disorders) | 1 (1) | 0 (0)
Nausea and vomiting (Gastrointestinal disorders) | 1 (1) | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ReShape Intragastric Balloon (N=21) | Control Arm (N=9)
nausea (Gastrointestinal disorders) | 21 (27) | 0 (0)
vomiting (Gastrointestinal disorders) | 18 (25) | 0 (0)
eructation (Gastrointestinal disorders) | 10 (11) | 0 (0)
abdominal pain upper (Gastrointestinal disorders) | 9 (10) | 0 (0)
gastroesophageal reflux disease (Gastrointestinal disorders) | 9 (12) | 0 (0)
abdominal discomfort (Gastrointestinal disorders) | 8 (8) | 0 (0)
dyspepsia (Gastrointestinal disorders) | 7 (7) | 0 (0)
gastric dilatation (Gastrointestinal disorders) | 7 (8) | 0 (0)
diarrhea (Gastrointestinal disorders) | 6 (7) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0)
constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
sinusitis (Infections and infestations) | 2 (2) | 2 (2)
upper respiratory tract infection (Infections and infestations) | 2 (3) | 0 (0)
urinary tract infection (Infections and infestations) | 2 (2) | 0 (0)
nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
dehydration (Metabolism and nutrition disorders) | 5 (5) | 0 (0)
back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 3 (3) | 0 (0)
migraine (Nervous system disorders) | 0 (0) | 1 (1)
anxiety (Psychiatric disorders) | 3 (3) | 0 (0)
vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Given the small sample size of this feasibility cohort, it was not expected to show significant effectiveness.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI shall furnish a copy of any proposed publication or disclosure at least 60 days prior to submission so that Sponsor may have the opportunity to protect its proprietary rights to information, inventions, or products developed under the Clinical Study. If such publication or disclosure contains Confidential Information, the PI agrees to remove such Confidential Information upon the Sponsor's request.